CLINICAL TRIAL: NCT02987673
Title: Effects of Mini/One Anastomosis Gastric Bypass (MGB/OAGB) and Sleeve Gastrectomy (LSG) on Lower Esophageal Sphincter (LES) Function. A Randomized Controlled Trial
Brief Title: MGB/OAGB and LSG Effects on Lower Esophageal Sphincter (LES) Function
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mario Musella MD (Other)
Responsible Party: Sponsor-Investigator, Mario Musella MD, Associate Professor of Surgery, Federico II University
Organization: Federico II University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MGB1
Record Dates: First submitted 2016-11-28; First posted 2016-12-09 (Estimated); Last update posted 2019-08-01 (Actual); Status verified 2019-07

CONDITIONS: Morbid Obesity; Gastroesophageal Reflux; Bariatric Surgery Candidate
Keywords: Mini/One anastomosis gastric bypass; Sleeve Gastrectomy; Gastro-esophageal sphincter function
MeSH Terms: conditions — Obesity, Morbid; Gastroesophageal Reflux

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mini/One anastomosis gastric bypass (Experimental): Execution of a laparoscopic mini/one anastomosis gastric bypass (MGB/OAGB)
  Interventions: Procedure: MGB/OAGB
- Laparoscopic sleeve gastrectomy (Active Comparator): Execution of a laparoscopic sleeve gastrectomy (LSG)
  Interventions: Procedure: LSG

INTERVENTIONS:
Procedure: MGB/OAGB
  Arms: Mini/One anastomosis gastric bypass
Procedure: LSG
  Arms: Laparoscopic sleeve gastrectomy

SUMMARY:
Background While several articles have reported about the effects of laparoscopic sleeve gastrectomy (LSG) on the lower esophageal sphincter (LES), to date, just one paper has discussed this issue with regard the Mini/One anastomosis gastric bypass (MGB/OAGB). This is expected to be the first randomized trial exploring and comparing these two interventions.

Setting "Federico II" University Hospital, Naples - ITALY.

Methods Fifty morbid obese patients are going to be studied. All patients presenting with a normal preoperative LES function will be randomly assigned to undergo LSG (arm 1 - 25 pts) or MGB (arm 2 - 25 pts). Patients undergo clinical assessment for reflux symptoms, and esophago-gastro-duodenoscopy (EGDS) plus high-resolution impedance manometry (HRiM) and 24-hour pH-impedance monitoring (MII-pH) before, two months and 1 year after both LSG or MGB/OAGB.

Objective Endpoint 1: Does this surgery affect the LES area function in both arm 1 or arm 2 patients determining a possible increase in gastroesophageal acid or non acid reflux? Endpoint 2: Does one between the two procedures outperform the other one in terms of eventual LES area modifications? Endpoint 3: In the case of a good performance of LSG or MGB/OAGB or both the procedures, is this to be primarily related to surgery per se or to weight loss?

ELIGIBILITY:
Inclusion Criteria:

* 80 morbid obese patients are going to be studied. All patients presenting with a normal preoperative LES function will be randomly assigned to undergo LSG (arm 1 - 40 pts) or MGB (arm 2 - 40 pts).-

Exclusion Criteria:

* Patients lost at follow up. Cancer patients at any stage.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2016-01; Primary Completion 2019-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Modifications in terms of LES function | 12 months
  Does this surgery affect the LES area function in both arm 1 or arm 2 patients determining a possible increase in gastroesophageal acid or non acid reflux? This will be measured by the numbers and the duration of both acidic and non acidic reflux measured by 24-hour pH-impedance monitoring (MII-pH)
Definition of the best procedure | 12 months
  Does one between the two procedures outperform the other one in terms of eventual LES area modifications? This will be measured in both procedures by the numbers and the duration of both acidic and non acidic reflux measured by 24-hour pH-impedance monitoring (MII-pH)

SECONDARY OUTCOMES:
Causes of eventual modifications of LES function in relationship with a specific surgical procedure | 6 months and 12 months
  In the case of a good performance of LSG or MGB/OAGB or both the procedures, is this to be primarily related to surgery per se or to weight loss? This will be evaluated in both procedures by the numbers and the duration of both acidic and non acidic reflux measured by 24-hour pH-impedance monitoring (MII-pH)
Causes of eventual modifications of LES function in relationship with weight loss | 6 months and 12 months
  In the case of a good performance of LSG or MGB/OAGB or both the procedures, is this to be primarily related to surgery per se or to weight loss? This will be evaluated in both procedures by the weight loss expressed as body mass index (BMI) points loss.

CONTACTS AND LOCATIONS:
Overall Officials: Mario Musella, MD, Principal Investigator — Federico II University
Locations (1):
- Advanced Biomedical Sciences Department - "Federico II" University, Naples, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Del Genio G, Tolone S, Limongelli P, Brusciano L, D'Alessandro A, Docimo G, Rossetti G, Silecchia G, Iannelli A, del Genio A, del Genio F, Docimo L. Sleeve gastrectomy and development of "de novo" gastroesophageal reflux. Obes Surg. 2014 Jan;24(1):71-7. doi: 10.1007/s11695-013-1046-4. PMID 24249251
- [Result] Melissas J, Braghetto I, Molina JC, Silecchia G, Iossa A, Iannelli A, Foletto M. Gastroesophageal Reflux Disease and Sleeve Gastrectomy. Obes Surg. 2015 Dec;25(12):2430-5. doi: 10.1007/s11695-015-1906-1. PMID 26428250
- [Result] Casella G, Soricelli E, Giannotti D, Collalti M, Maselli R, Genco A, Redler A, Basso N. Long-term results after laparoscopic sleeve gastrectomy in a large monocentric series. Surg Obes Relat Dis. 2016 May;12(4):757-762. doi: 10.1016/j.soard.2015.09.028. Epub 2015 Oct 1. PMID 26806727
- [Result] Tolone S, Cristiano S, Savarino E, Lucido FS, Fico DI, Docimo L. Effects of omega-loop bypass on esophagogastric junction function. Surg Obes Relat Dis. 2016 Jan;12(1):62-9. doi: 10.1016/j.soard.2015.03.011. Epub 2015 Mar 27. PMID 25979206